CLINICAL TRIAL: NCT01422889
Title: A U.S. Post-Approval Study of the ION™ Paclitaxel-Eluting Platinum Chromium Coronary Stent System
Brief Title: ION US Post-Approval Study
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: S2065
Record Dates: First submitted 2011-08-22; First posted 2011-08-25 (Estimated); Results first posted 2015-03-20 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-01

CONDITIONS: Atherosclerosis; Coronary Artery Disease
Keywords: Atherosclerosis; Coronary Artery Disease
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ION Registry: The ION Registry population was designed to collect real world safety and clinical outcomes data. There were 1120 subjects were enrolled, however 9 subjects did not receive a study stent therefore 1111 subjects were eligible for follow up.
  Interventions: Device: ION™ Coronary Stent System

INTERVENTIONS:
Device: ION™ Coronary Stent System — This study is intended to evaluate the ION™ Paclitaxel-Eluting Platinum Chromium Coronary Stent System across a range of institutions and physician users to observe and assess subject outcomes and technology performance in a real-world setting.

SUMMARY:
The purpose of this study is to compile real-world clinical outcomes data for the ION™ Paclitaxel-Eluting Platinum Chromium Coronary Stent System in routine clinical practice.

DETAILED DESCRIPTION:
The ION™ stent is the third-generation Boston Scientific (BSC) paclitaxel-eluting coronary stent. It is designed for improved performance specific to deliverability and radio-opacity while maintaining a similar drug release profile of the TAXUS Express and TAXUS Liberté stents. Following PMA approval from the FDA for the ION™ Paclitaxel-Eluting Platinum Chromium Coronary Stent System the ION US Post-Approval study will compile real-world clinical outcomes data for the ION™ Paclitaxel-Eluting Platinum Chromium Coronary Stent System in routine clinical practice. Post-approval studies of drug-eluting stents (DES) provide an opportunity to observe and assess patient outcomes and technology performance in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

Consented subjects receiving one or more ION(TM)Coronary Stents

Exclusion Criteria:

Subjects not clinically indicated to receive an ION (TM)Coronary Stent

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consented subjects admitted to the cardiac catheterization laboratory for percutaneous transluminal coronary angioplasty and who are eligible to receive an ION™ Paclitaxel-Eluting Platinum Chromium Coronary Stent.
Sampling Method: Non-Probability Sample
Enrollment: 1120 (Actual)
Dates: Start 2011-09; Primary Completion 2013-06 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis A Cannon, MD, Principal Investigator — Northern Michigan Hospital; Carey D Kimmelstiel, MD, Principal Investigator — Tufts Medical Center
Locations (40):
- United States (40):
  - NEA Baptist Memorial Hospital, Jonesboro, Arkansas
  - St. Bernard's Medical Center, Jonesboro, Arkansas
  - Bakersfield Memorial Hospital, Bakersfield, California
  - Alvarado Hospital, San Diego, California
  - Northside Hospital and Heart Institute, St. Petersburg, Florida
  - University Community Hospital, Tampa, Florida
  - Redmond Regional Medical Center, Rome, Georgia
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Krannert Institute of Cardiology, Indianapolis, Indiana
  - Indiana Heart Hospital, Indianapolis, Indiana
  - Iowa Heart Center, West Des Moines, Iowa
  - King's Daughters Medical Center - Kentucky Heart Inst, Ashland, Kentucky
  - Maine Medical Center, Portland, Maine
  - Union Memorial Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Sparrow Health System - Sparrow Hospital, Lansing, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - Lakeland Hospitals at St. Joseph, Saint Joseph, Michigan
  - Memorial Hospital at Gulfport, Gulfport, Mississippi
  - Freeman West Hospital, Joplin, Missouri
  - Our Lady of Lourdes Medical Center, Haddon Heights, New Jersey
  - Jersey Shore University Medical Center, Sea Girt, New Jersey
  - St. Joseph's Hospital Health Center, Liverpool, New York
  - St. Elizabeth Medical Center, Utica, New York
  - Wake Medical Center, Raleigh, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Mercy St. Vincent Medical Center, Toledo, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - St. Mary Medical Center, Yardley, Pennsylvania
  - Sisters of Charity Providence Hospital, Columbia, South Carolina
  - Grand Strand Regional Medical Center, Myrtle Beach, South Carolina
  - Regional Hospital, Jackson, Tennessee
  - Centennial Medical Center, Nashville, Tennessee
  - Baylor Heart & Vascular Hospital, Dallas, Texas
  - CRSTI/Medical City Dallas, Dallas, Texas
  - Kingwood Medical Center Hospital, Kingwood, Texas
  - Methodist Texsan Hospital, San Antonio, Texas
  - Meriter Hospital, Inc., Madison, Wisconsin
  - CaRE Foundation, Inc., Wausau, Wisconsin

REFERENCES:
- [Result] Cannon L, Kimmelstiel CD, Kellett M, White A, Hill R, Grady T, Myers PR, Underwood P, Dawkins KD. One-year real-world outcomes following implantation of the ION paclitaxel-eluting platinum chromium coronary stent in routine clinical practice: Primary endpoint results of the ION U.S. post-approval registry [abstract]. J Am Coll Cardiol. 2013; 62 (18 SUPPL. 1): B58
- [Result] Kimmelstiel CD, Cannon LA, Jobe RL, Stoler R, Pow T, Ganim R, Kayser R, Allocco DJ, Dawkins KD. Two-Year "Real-World" Outcomes Following Implantation of the ION™ Paclitaxel-Eluting Platinum Chromium Coronary Stent in Routine Clinical Practice: Results From the ION U.S. Post-Approval Registry. Presented at: The Transcatheter and Cardiovascular Therapeutics Annual Meeting 2014; Washington, D.C, USA. September 13 - 17, 2014.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment began on 19 September 2011 and was completed on 24 April 2012.
Groups:
- ION Registry: The ION Registry population consists of 1111 subjects that were enrolled and received a study stent.
Period: Overall Study
Arm/Group | ION Registry
Started | 1120
Completed | 1111 (9 subjects did not receive a study stent therefore 1111 subjects were eligible for follow up.)
Not Completed | 9
Not completed — No Data Entered for Study Stent | 9

BASELINE CHARACTERISTICS:
Population: Subjects that recevied at least one study stent
Groups:
- ION Registry: The ION Registry population contains 1120 enrolled subjects with 1111 eligible for analysis. Subjects eligible for analysis includes subjects with at least one study stent implanted.
Arm/Group | ION Registry
Number analyzed (Participants) | 1111
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 330
  Male | 781
Region of Enrollment [Number; unit: participants]
  United States | 1111
Cardiac Risk Factors [Number; unit: participants] — The same participant may be included in more than one category therefore the number of participants does not equal the total number of participants in the group.
  participants
    Diabetes | 376
    Current Smoker | 275
    Hypertension | 905
    Hyperlipidemia | 869
    Unstable Angina | 485
    Prior PCI | 522
Lesion Characteristics [Number; unit: participants] — The same participant may be included in more than one category therefore the number of participants does not equal the total number of participants in the group.
  participants
    RVD<=2.5mm | 387
    Long Lesions (>=28mm) | 235
    Bifurcation | 116
Lesion Characteristics:Lesion Based [Number; unit: Lesions] — N=1111 subjects; N=1562 Lesions
  Lesions
    Culprit for STEMI | 108
    Severe Calcification | 79

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Death or Myocardial Infarction (CD/MI)
Description: Cardiac Death or myocardial infarction (CD/MI) in the ION registry population. For the protocol specified primary endpoint analysis including data pooled from the PERSEUS SV, PERSEUS WH and TE Prove patient populations please see the citations.
Time Frame: 12 Months
Population: There were 83 subjects not evaluable for 12-month cardiac events (No follow-up ≥ 335 days and events-free within 365-day) leaving a total of 1028 subjects evaluated for 12 month CD/MI.
Measure: Number; unit: percentage of paricipants
Groups:
- ION Registry: The ION Registry includes the 1111 enrolled subjects that received a study stent.
Arm/Group | ION Registry
Number analyzed (Participants) | 1028
percentage of paricipants | 2.2
Statistical Analysis 1: Comparison: ION Registry; 2.2% (23/1028) of ION Registry subjects experienced CD/MI related to the ION stent at 12 months; Test type: Superiority or Other; A p-value was not calculated for the ION Registry 12 month cardiac events. For the protocol specified primary endpoint analysis including data pooled from the PERSEUS SV, PERSEUS WH and TE Prove patient populations please see the citations; percentage = 2.2

2. Secondary Outcome: Stent Thrombosis
Description: Academic Research Consortium (ARC) defined (definite/probable) stent thrombosis (ST) in the ION registry population. For the protocol specified secondary endpoint analysis including data pooled from the PERSEUS SV, PERSEUS WH and TE Prove patient populations please see the citations.
Time Frame: Annually, after the first year, through 2 years.
Population: There were 57 subjects not evaluable for 2-year cardiac events (No follow-up ≥ 700 days and events-free within 730-day) leaving a total of 1054 subjects evaluated for ARC ST Definite/Probable.
Measure: Number; unit: percentage of participants
Arm/Group | ION Registry
Number analyzed (Participants) | 1054
percentage of participants | 2.6
Statistical Analysis 1: Comparison: ION Registry; 2.6% (27/1054) of ION Registry subjects experienced ARC ST Definite/Probable related to the ION stent at 2 years; Test type: Superiority or Other; A p-value was not calculated for the ION Registry 2 year cardiac events. For the protocol specified secondary endpoint analysis including data pooled from the PERSEUS SV, PERSEUS WH and TE Prove patient populations please see the citations; percentage = 2.6

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- ION Registry: The ION Registry population will contain the first 1115 consecutive, consenting patients
Arm/Group | ION Registry
Serious Adverse Events (participants affected / at risk) | 324/1111
Other Adverse Events (participants affected / at risk) | 0/1111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ION Registry (N=1111)
Angina Pectoris (Cardiac disorders) | 59 (70)
Angina Unstable (Cardiac disorders) | 23 (31)
Acute Myocardial Infarction (Cardiac disorders) | 27 (27)
Cardiac Congestive Failure (Cardiac disorders) | 23 (26)
Coronary artery thrombosis (Cardiac disorders) | 15 (18)
Myocardial Infarction (Cardiac disorders) | 17 (17)
Atrial Fibriliation (Cardiac disorders) | 14 (17)
Coronary artery disease (Cardiac disorders) | 13 (14)
Cardiac arrest (Cardiac disorders) | 7 (7)
Acute Coronary System (Cardiac disorders) | 5 (5)
Cardiac failure (Cardiac disorders) | 4 (4)
Coronary artery stenosis (Cardiac disorders) | 4 (4)
Ventricular fibrillation (Cardiac disorders) | 4 (4)
Atrial flutter (Cardiac disorders) | 3 (4)
Cardiac failure chronic (Cardiac disorders) | 3 (4)
Cardiogenic shock (Cardiac disorders) | 3 (4)
Ischaemic cardiomyopathy (Cardiac disorders) | 3 (4)
Ventricular tachycardia (Cardiac disorders) | 2 (4)
Cardiomyopathy (Cardiac disorders) | 3 (3)
Arrhythmia supraventricular (Cardiac disorders) | 2 (2)
Atrioventricular block (Cardiac disorders) | 2 (2)
Coronary artery dissection (Cardiac disorders) | 2 (2)
Pericarditis (Cardiac disorders) | 2 (2)
Sick sinus syndrome (Cardiac disorders) | 2 (2)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1)
Chronotropic incompetence (Cardiac disorders) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Sinus arrest (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Pneumonia (Infections and infestations) | 18 (22)
Urinary tract infection (Infections and infestations) | 10 (10)
Sepsis (Infections and infestations) | 5 (5)
Diverticulitis (Infections and infestations) | 4 (5)
Bronchitis (Infections and infestations) | 3 (3)
Cellulitis (Infections and infestations) | 3 (3)
Abscess (Infections and infestations) | 2 (2)
Appendicitis (Infections and infestations) | 2 (2)
Gastroenteritis (Infections and infestations) | 2 (2)
Arthritis bacterial (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Gangrene (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Infected skin ulcer (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Osteomyelitis acute (Infections and infestations) | 1 (1)
Periorbital abscess (Infections and infestations) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Non-cardiac chest pain (General disorders) | 35 (46)
Chest pain (General disorders) | 6 (6)
Chest discomfort (General disorders) | 3 (3)
Pyrexia (General disorders) | 3 (3)
Asthenia (General disorders) | 1 (1)
Catheter site haematoma (General disorders) | 1 (1)
Hernia obstructive (General disorders) | 1 (1)
Sudden cardiac death (General disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 11 (12)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Colonic polyp (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1)
Epiploic appendagitis (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Intestional perforation (Gastrointestinal disorders) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 4 (6)
Peripheral vascular disorder (Vascular disorders) | 4 (5)
Aortic stenosis (Vascular disorders) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Femoral arterial stenosis (Vascular disorders) | 2 (2)
Intermittent claudication (Vascular disorders) | 2 (2)
Aortic aneurysm (Vascular disorders) | 1 (1)
Arterial haemorrhage (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Iliac artery embolism (Vascular disorders) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 1 (1)
Leriche syndrome (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1)
Syncope (Nervous system disorders) | 8 (8)
Cerebrovascular accident (Nervous system disorders) | 6 (6)
Carotid artery stenosis (Nervous system disorders) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 2 (2)
Ataxia (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Migrane (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 14 (17)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2 (2)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 7 (7)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 2 (2)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1)
Device malfunction (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1)
Renal injury (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Renal failure (Renal and urinary disorders) | 4 (4)
Renal failure acute (Renal and urinary disorders) | 3 (3)
Renal failure chronic (Renal and urinary disorders) | 3 (3)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 1 (1)
Renal disorder (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Vaginal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Hepatic artery stenosis (Hepatobiliary disorders) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1)
Hepatic congestion (Hepatobiliary disorders) | 1 (1)
Ischaemic hepatitis (Hepatobiliary disorders) | 1 (1)
Cardiac stress test abnormal (Investigations) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1)
Heart rate increased (Investigations) | 1 (1)
International normalized ratio increased (Investigations) | 1 (1)
Intervertebral disc protusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Cataract (Eye disorders) | 2 (2)
Conjunctival haemorrhage (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin plaque (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Bipolar I disorder (Psychiatric disorders) | 1 (1)
Deperession (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1)
Congenital coronary artery malformation (Congenital, familial and genetic disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Cardiac pacemaker battery replacement (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less